CLINICAL TRIAL: NCT03030222
Title: Empagliflozin Evaluation by Measuring Impact on Hemodynamics in Patients With Heart Failure
Brief Title: Empagliflozin Impact on Hemodynamics in Patients With Heart Failure
Acronym: EMBRACE-HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Saint Luke's Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1245.129
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Results first posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Heart Failure
Keywords: heart failure; empagliflozin; Sodium-glucose Cotransporter-2 (SGLT2) Inhibitors
MeSH Terms: conditions — Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin (Active Comparator): Empagliflozin 10 mg tab, once daily, for 12 weeks
  Interventions: Drug: Empagliflozin 10 mg Tab
- Placebo (Placebo Comparator): Empagliflozin matching placebo oral tablet, once daily for 12 weeks
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Empagliflozin 10 mg Tab — Empagliflozin 10 mg Tab
  Other Names: Jardiance
  Arms: Empagliflozin
Drug: Placebo Oral Tablet — Empagliflozin matching placebo
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The primary purpose of this trial is to evaluate the impact of empagliflozin, as compared with placebo, on hemodynamic parameters (pulmonary artery diastolic pressure) in patients with heart failure (reduced or preserved ejection fraction, ischemic or non-ischemic etiology) who already have a CardioMEMs device (a wireless hemodynamic monitoring system) implanted for non-study related clinical reasons.

DETAILED DESCRIPTION:
A 12-week randomized, double-blind, placebo-controlled trial to explore the effects of once-daily empagliflozin 10 mg on hemodynamic parameters (pulmonary artery pressures) in patients with heart failure (reduced or preserved ejection fraction, ischemic or non-ischemic etiology) who already have a CardioMEMs device implanted for non-study related clinical reasons.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of heart failure (for at least 16 weeks prior to the screening visit) with either preserved (LVEF>40%) or reduced systolic function (LVEF≤40%), due to either ischemic or non-ischemic etiology, documented by an imaging modality (echocardiography, nuclear imaging, LV angiography, magnetic resonance imaging) within the past 24 months.
2. No major change in diuretic management for 48 hours prior to screening visit or 48 hours prior to randomization visit (major change defined by doubling of diuretic dose or addition of another diuretic medication)
3. New York Heart Association (NYHA) class II, III or IV heart failure symptoms at the screening and randomization visit
4. Presence of previously (≥ 2 weeks prior to screening visit) implanted CardioMEMs pulmonary artery pressure monitor for a clinical indication unrelated to the study.
5. Pulmonary artery diastolic pressure ≥ 12 mmHg at the time of the screening visit (last measurement available prior to the screening visit).
6. Ability to provide informed consent prior to initiating screening visit procedures

Exclusion Criteria:

1. Decompensated heart failure (hospitalization for heart failure within the 2 weeks prior to screening) or between screening and randomization
2. History of type 1 diabetes
3. Major change in diuretic management during 48 hours prior to screening visit or 48 hours prior to randomization visit. (major change defined by doubling of diuretic dose or addition of another diuretic medications)
4. Significant variability in baseline pulmonary artery diastolic pressures during screening period. Defined as changes greater than +/- 6 mmHg from average pulmonary artery diastolic pressure during week 1 of the screening phase and average pulmonary artery diastolic pressure during week 2 of the screening phase for those patients with an average baseline pulmonary artery diastolic pressure during week 1 of the screening phase of <30 mmHg. If the average baseline pulmonary artery diastolic pressure during week 1 of the screening phase is ≥30 mmHg, then ≥20% relative change in average pulmonary diastolic pressure between week 1 and week 2 of the screening phase will be used to define significant variability.
5. Initiation of hydralazine, long-acting nitrates, beta blockers, angiotensin-converting enzyme inhibitors (ACEIs) , angiotensin II receptor blockers (ARBs) or valsartan/sacubitril in the prior 4 weeks prior to screening
6. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 at the screening visit
7. Admission for an acute coronary syndrome (ST-elevation myocardial infarction, non-ST-elevation myocardial infarction, or unstable angina), percutaneous coronary intervention, or cardiac surgery within 30 days prior to the screening visit.
8. Implantation of cardiac resynchronization therapy (CRT) device within the previous 90 days.
9. Implantation of the CardioMEMs device within the past 2 weeks.
10. Planned cardiovascular revascularization (percutaneous intervention or surgical) or major cardiac surgery (coronary artery bypass grafting, valve replacement, ventricular assist device, cardiac transplantation, or any other surgery requiring thoracotomy), or planned implantation of cardiac resynchronization therapy (CRT) device within the 90 days after the screening visit.
11. Participation in any interventional clinical trial (with an investigational drug or device) that is not an observational registry within the 4 weeks prior to the screening visit.
12. History of hypersensitivity to empagliflozin
13. For women of child-bearing potential: Current or planned pregnancy or currently lactating
14. Life expectancy <1 year at the screening visit
15. Patients who are volume depleted based upon physical examination at the time of the screening or randomization visit
16. Pulmonary artery diastolic pressure < 12 mmHg at the time of the screening visit (average of last four measurements available prior to the screening visit).
17. Patients currently being treated with any SGLT-2 inhibitor (dapagliflozin, canagliflozin, empagliflozin) or having received treatment with any SGLT-2 inhibitor within the 8 weeks prior to the screening visit
18. Average supine systolic BP <90 mmHg at the screening or randomization visit
19. Current documented history of bladder cancer
20. Active Gross Hematuria
21. Heart failure due to restrictive cardiomyopathy, active myocarditis, constrictive pericarditis, severe stenotic valve disease, and hypertrophic obstructive cardiomyopathy (HOCM).
22. History of heart transplant.
23. Patients on heart transplant list as 1a and 1b status

Ages: 19 Years to 119 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Kosiborod, MD, Study Chair — Saint Luke's Mid America Heart Institute
Locations (10):
- United States (10):
  - University of Southern California, Los Angeles, California
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - NorthShore University Health System Research Institute, Evanston, Illinois
  - CentraCare Heart and Vascular Center, Saint Cloud, Minnesota
  - St. Francis Hospital, Roslyn, New York
  - Ohio State University, Columbus, Ohio
  - Sanford Research, Sioux Falls, South Dakota
  - Austin Heart Clinical Research, Austin, Texas
  - Baylor College of Medicine, Houston, Texas
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nassif ME, Qintar M, Windsor SL, Jermyn R, Shavelle DM, Tang F, Lamba S, Bhatt K, Brush J, Civitello A, Gordon R, Jonsson O, Lampert B, Pelzel J, Kosiborod MN. Empagliflozin Effects on Pulmonary Artery Pressure in Patients With Heart Failure: Results From the EMBRACE-HF Trial. Circulation. 2021 Apr 27;143(17):1673-1686. doi: 10.1161/CIRCULATIONAHA.120.052503. Epub 2021 Feb 8. PMID 33550815
- [Derived] Nassif ME, Spertus JA, Tang F, Windsor SL, Jones P, Thomas M, Khariton Y, Brush J, Gordon RA, Jermyn R, Jonsson O, Lamba S, Shavelle DM, Kosiborod MN. Association Between Change in Ambulatory Hemodynamic Pressures and Symptoms of Heart Failure. Circ Heart Fail. 2021 Nov;14(11):e008446. doi: 10.1161/CIRCHEARTFAILURE.121.008446. Epub 2021 Oct 26. No abstract available. PMID 34696602
- [Derived] Nassif ME, Kosiborod M. Effects of sodium glucose cotransporter type 2 inhibitors on heart failure. Diabetes Obes Metab. 2019 Apr;21 Suppl 2:19-23. doi: 10.1111/dom.13678. PMID 31081589
- See also: Empagliflozin information — https://druginfo.nlm.nih.gov/drugportal/name/empagliflozin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Empagliflozin | Placebo
Started | 33 | 32
Completed | 33 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Empagliflozin | Placebo | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (12.0) | 62.9 (13.3) | 66.2 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 21 | 20 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 7 | 12
  White | 27 | 23 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 33 | 32 | 65
Duration of Heart Failure [Mean (Standard Deviation); unit: years] | 5.4 (5.7) | 7.2 (5.5) | 6.3 (5.6)
Prior hospitalization for heart failure [Count of Participants; unit: Participants] | 29 | 28 | 57
Time since last hospitalization for heart failure [Mean (Standard Deviation); unit: years] | 1.3 (0.9) | 1.5 (1.4) | 1.4 (1.2)
Ejection fraction [Mean (Standard Deviation); unit: %] | 46.7 (14.9) | 40.7 (17.2) | 43.7 (16.2)
Ischemic heart disease [Count of Participants; unit: Participants] | 13 | 10 | 23
Type 2 Diabetes [Count of Participants; unit: Participants] | 18 | 16 | 34
Atrial Fibrillation [Count of Participants; unit: Participants] | 20 | 17 | 37
Implantable cardioverter defibrillator (ICD) [Count of Participants; unit: Participants] | 15 | 21 | 36
Cardiac resynchronization therapy (CRT) [Count of Participants; unit: Participants] | 13 | 8 | 21
Pulmonary Artery Diastolic Pressure [Mean (Standard Deviation); unit: mm Hg] | 23.3 (6.9) | 20.5 (5.7) | 21.9 (6.4)
Angiotensin-converting enzyme inhibitor / Angiotensin II receptor blocker (ACEI/ARB) [Count of Participants; unit: Participants] | 11 | 8 | 19
Angiotensin receptor-neprilysin inhibitor (ARNI) [Count of Participants; unit: Participants] | 13 | 17 | 30
Beta blockers [Count of Participants; unit: Participants] | 29 | 29 | 58
Hydralazine [Count of Participants; unit: Participants] | 7 | 3 | 10
Long-acting nitrates [Count of Participants; unit: Participants] | 15 | 9 | 24
Mineralocorticoid receptor antagonist (MRA) [Count of Participants; unit: Participants] | 9 | 20 | 29
Loop diuretics [Count of Participants; unit: Participants] | 31 | 32 | 63
Digoxin [Count of Participants; unit: Participants] | 6 | 3 | 9
Lipid lowering agent [Count of Participants; unit: Participants] | 27 | 23 | 50
Anticoagulant agent [Count of Participants; unit: Participants] | 16 | 13 | 29
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 33.5 [28.6 to 39.5] | 33.8 [29.4 to 40.0] | 33.5 [28.8 to 40.0]
Heart rate [Mean (Standard Deviation); unit: bpm] | 70.1 (10.2) | 72.6 (9.8) | 71.3 (10)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 128.3 (19.1) | 120.7 (20.3) | 124.5 (19.9)
N-terminal pro b-type natriuretic peptide (NT-proBNP) [Median (Inter-Quartile Range); unit: pg/mL] | 865.5 [311.0 to 1982.5] | 563.5 [153.0 to 1964.0] | 637.0 [249.5 to 1964.0]
Brain natriuretic peptide (BNP) [Median (Inter-Quartile Range); unit: pg/mL] | 140.0 [85.0 to 286.0] | 129.0 [51.0 to 378.5] | 140 [57.0 to 293.0]
Estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 51.2 (19.7) | 62.7 (25.5) | 56.9 (23.3)
Urine Albumin/Creatinine Ratio [Mean (Standard Deviation); unit: mg/g] | 101.9 (187.4) | 201.6 (688.2) | 149.3 (491.1)
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of hemoglobin] | 6.4 (1.3) | 6.9 (1.9) | 6.6 (1.6)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 13.3 (2.1) | 12.5 (1.6) | 12.9 (1.9)
New York Heart Association (NYHA) Class II [Count of Participants; unit: Participants] — Doctors usually classify patients' heart failure according to the severity of their symptoms. The most commonly used classification system is the New York Heart Association (NYHA) Functional Classification. It places patients in one of four categories based on how much they are limited during physical activity. NYHA Class II means the patient has been classified as having slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  Participants | 14 | 16 | 30
New York Heart Association (NYHA) Class III [Count of Participants; unit: Participants] — Doctors usually classify patients' heart failure according to the severity of their symptoms. The most commonly used classification system is the New York Heart Association (NYHA) Functional Classification. It places patients in one of four categories based on how much they are limited during physical activity. NYHA Class III indicates the patient has been classified as having Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Participants | 18 | 16 | 34
Kansas City Cardiomyopathy Questionnaire - Overall Summary Score (KCCQ-OS) [Mean (Standard Deviation); unit: points] — The KCCQ is a disease-specific health status instrument composed of 23 items that quantifies the domains of physical limitations, symptoms, self-efficacy, social limitation and quality of life from heart failure. Scores range from 0-100, in which higher scores reflect better health status.
  points | 60.5 (16.9) | 61.1 (27.2) | 60.8 (22.4)
Kansas City Cardiomyopathy Questionnaire - Clinical Summary Score (KCCQ-CS) [Mean (Standard Deviation); unit: points] — The KCCQ is a disease-specific health status instrument composed of 23 items that quantifies the domains of physical limitations, symptoms, self-efficacy, social limitation and quality of life from heart failure. Scores range from 0-100, in which higher scores reflect better health status.
  points | 60.2 (18.7) | 64.6 (26.4) | 62.4 (22.8)
6-minute walk distance [Median (Inter-Quartile Range); unit: meters] | 237.7 [158.5 to 259.1] | 232.1 [181.4 to 330.7] | 233.2 [170.7 to 304.8]
Insulin (among patients with type 2 diabetes) [Count of Participants; unit: Participants] — Population: Insulin use among patients with type 2 diabetes.
  Participants
    number analyzed (Participants) | 18 | 16 | 34
    (all) | 11 | 11 | 22
Glucagon-like peptide-1 receptor agonist (GLP-1 RA )(among patients with type 2 diabetes) [Count of Participants; unit: Participants] — Population: GLP-1RA use among patients with type 2 diabetes.
  Participants
    number analyzed (Participants) | 18 | 16 | 34
    (all) | 3 | 4 | 7
Dipeptidyl-peptidase 4 (DPP4) inhibitor (among patients with type 2 diabetes) [Count of Participants; unit: Participants] — Population: DPP4-inhibitor use among patients with type 2 diabetes.
  Participants
    number analyzed (Participants) | 18 | 16 | 34
    (all) | 2 | 2 | 4
Sulfonylurea (among patients with type 2 diabetes) [Count of Participants; unit: Participants] — Population: Sulfonylurea use among patients with type 2 diabetes.
  Participants
    number analyzed (Participants) | 18 | 16 | 34
    (all) | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Pulmonary Artery Diastolic Pressure From Baseline to End of Treatment Period (Defined as Average of Pulmonary Artery Diastolic Pressure Measurements Between Weeks 8-12) Between Empagliflozin and Placebo
Description: Change in pulmonary artery diastolic pressure from baseline to end of treatment period (defined as average of pulmonary artery diastolic pressure measurements between weeks 8-12) between empagliflozin and placebo
Time Frame: Baseline to average between Weeks 8-12
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 33 | 32
mm Hg | 20.7 [19.6 to 21.7] | 22.2 [21.1 to 23.2]

2. Secondary Outcome: Change From Baseline in Pulmonary Artery Diastolic Pressure at Each Interim Timepoint (Wks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11,12) Between Empagliflozin and Placebo.
Description: Change from baseline in pulmonary artery diastolic pressure at each interim timepoint (wks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11,12) between empagliflozin and placebo.
Time Frame: Baseline to Weeks 1-12
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 33 | 32
mm Hg
  Pulmonary artery diastolic pressure - Week 0 | 21.2 [20.4 to 22.1] | 21.4 [20.5 to 22.2]
  Pulmonary artery diastolic pressure - Week 1 | 21.2 [20.4 to 21.9] | 21.5 [20.7 to 22.3]
  Pulmonary artery diastolic pressure - Week 2 | 21.1 [20.3 to 21.9] | 21.7 [20.9 to 22.4]
  Pulmonary artery diastolic pressure - Week 3 | 21.1 [20.2 to 21.9] | 21.8 [20.9 to 22.6]
  Pulmonary artery diastolic pressure - Week 4 | 21.0 [20.1 to 22.0] | 21.9 [21.0 to 22.8]
  Pulmonary artery diastolic pressure - Week 5 | 21.0 [20.1 to 22.0] | 22.0 [21.0 to 23.0]
  Pulmonary artery diastolic pressure - Week 6 | 21.0 [20.0 to 22] | 22.1 [21.1 to 23.1]
  Pulmonary artery diastolic pressure - Week 7 | 21.0 [19.9 to 22.0] | 22.1 [21.1 to 23.2]
  Pulmonary artery diastolic pressure - Week 8 | 21.0 [19.8 to 22.0] | 22.2 [21.1 to 23.2]
  Pulmonary artery diastolic pressure - Week 9 | 20.8 [19.7 to 21.9] | 22.2 [21.1 to 23.3]
  Pulmonary artery diastolic pressure - Week 10 | 20.7 [19.6 to 21.8] | 22.2 [21.1 to 23.3]
  Pulmonary artery diastolic pressure - Week 11 | 20.5 [19.5 to 21.6] | 22.2 [21.0 to 23.3]
  Pulmonary artery diastolic pressure - Week 12 | 20.4 [19.2 to 21.6] | 22.1 [20.9 to 23.3]

3. Secondary Outcome: Change in Pulmonary Artery Systolic Pressure From Baseline to End of Treatment Period (Week 12) Between Empagliflozin and Placebo.
Description: Change in pulmonary artery systolic pressure from baseline to end of treatment period (week 12) between empagliflozin and placebo.
Time Frame: Baseline to Week 12
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 33 | 32
mm Hg | 20.4 [19.2 to 21.6] | 22.1 [20.9 to 23.3]

4. Secondary Outcome: Change From Baseline in Pulmonary Artery Systolic Pressure at Each Interim Time Point (Wks 1, 2, 3, 4, 5, 6, 7, 8, 9,10,11,12) Between Empagliflozin and Placebo.
Description: Change from baseline in pulmonary artery systolic pressure at each interim time point (wks 1, 2, 3, 4, 5, 6, 7, 8, 9,10,11,12) between empagliflozin and placebo.
Time Frame: Baseline to Weeks 1-12
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 33 | 32
mm Hg
  Pulmonary artery systolic pressure - Week 0 | 44.1 [42.6 to 45.6] | 43.9 [42.4 to 45.3]
  Pulmonary artery systolic pressure - Week 1 | 44.1 [42.8 to 45.4] | 44.0 [42.7 to 45.2]
  Pulmonary artery systolic pressure - Week 2 | 44.1 [42.8 to 45.4] | 44.1 [42.8 to 45.3]
  Pulmonary artery systolic pressure - Week 3 | 44.1 [42.6 to 45.5] | 44.2 [42.7 to 45.6]
  Pulmonary artery systolic pressure - Week 4 | 44.0 [42.5 to 45.6] | 44.3 [42.7 to 45.8]
  Pulmonary artery systolic pressure - Week 5 | 44.0 [42.3 to 45.6] | 44.4 [42.8 to 46.0]
  Pulmonary artery systolic pressure - Week 6 | 44.0 [42.2 to 45.6] | 44.6 [42.9 to 46.3]
  Pulmonary artery systolic pressure - Week 7 | 43.8 [42.0 to 45.6] | 44.7 [42.9 to 46.5]
  Pulmonary artery systolic pressure - Week 8 | 43.7 [41.8 to 45.6] | 44.8 [42.9 to 46.8]
  Pulmonary artery systolic pressure - Week 9 | 43.6 [41.6 to 45.5] | 44.9 [42.9 to 46.9]
  Pulmonary artery systolic pressure - Week 10 | 43.4 [41.5 to 45.3] | 44.9 [43.0 to 46.9]
  Pulmonary artery systolic pressure - Week 11 | 43.3 [41.3 to 45.2] | 44.9 [43.0 to 46.9]
  Pulmonary artery systolic pressure - Week 12 | 43.1 [41.0 to 45.1] | 44.9 [42.8 to 46.9]

5. Secondary Outcome: Change in Mean Pulmonary Artery Pressure From Baseline to End of Treatment Period (Week 12) Between Empagliflozin and Placebo.
Description: Change in mean pulmonary artery pressure from baseline to end of treatment period (week 12) between empagliflozin and placebo.
Time Frame: Baseline to Week 12
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 33 | 32
mm Hg | 29.3 [27.9 to 30.8] | 31.1 [29.6 to 32.5]

6. Secondary Outcome: Change From Baseline in Mean Pulmonary Artery Pressure at Each Interim Time Point (Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12) Between Empagliflozin and Placebo.
Description: Change from baseline in mean pulmonary artery pressure at each interim time point (weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12) between empagliflozin and placebo.
Time Frame: Baseline to Weeks 1-12
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 33 | 32
mm Hg
  Pulmonary artery pressure - Week 0 | 30.1 [29.0 to 31.2] | 30.1 [29.0 to 31.2]
  Pulmonary artery pressure - Week 1 | 30.1 [29.1 to 31.1] | 30.2 [29.2 to 31.2]
  Pulmonary artery pressure - Week 2 | 30.1 [29.1 to 31.0] | 30.4 [29.4 to 31.4]
  Pulmonary artery pressure - Week 3 | 30.0 [29.0 to 31.1] | 30.5 [29.5 to 31.6]
  Pulmonary artery pressure - Week 4 | 30.0 [28.9 to 31.2] | 30.7 [29.5 to 31.8]
  Pulmonary artery pressure - Week 5 | 30.0 [28.8 to 31.2] | 30.8 [29.6 to 32.0]
  Pulmonary artery pressure - Week 6 | 30.0 [28.7 to 31.2] | 30.9 [29.7 to 32.2]
  Pulmonary artery pressure - Week 7 | 29.9 [28.6 to 31.2] | 31.0 [29.7 to 32.3]
  Pulmonary artery pressure - Week 8 | 29.9 [28.5 to 31.2] | 31.1 [29.7 to 32.4]
  Pulmonary artery pressure - Week 9 | 29.8 [28.4 to 31.1] | 31.1 [29.7 to 32.5]
  Pulmonary artery pressure - Week 10 | 29.6 [28.2 to 31] | 31.1 [29.8 to 32.5]
  Pulmonary artery pressure - Week 11 | 29.5 [28.1 to 30.8] | 31.1 [29.7 to 32.5]
  Pulmonary artery pressure - Week 12 | 29.3 [27.9 to 30.8] | 31.1 [29.6 to 32.5]

7. Secondary Outcome: Change in Heart Failure Related Quality of Life, Using the Kansas City Cardiomyopathy Questionnaire Overall Summary Score (KCCQ-OS) From Baseline to Follow-up (Defines as Average of Measurements at 6 and 12 Weeks) Between Empagliflozin and Placebo.
Description: The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a disease-specific health status instrument composed of 23 items that quantifies the domains of physical limitations, symptoms, self-efficacy, social limitation and quality of life from heart failure. Scores range from 0-100, in which higher scores reflect better health status. For the Kansas City Cardiomyopathy Questionnaire Overall Summary Score KCCQ-OS, a small but clinically meaningful change is considered to be ≥ 5 points.
Time Frame: Baseline to Week 6 and Week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 33 | 32
score on a scale
  Kansas City Cardiomyopathy Questionnaire Overall Summary Score (KCCQ-OS) score - 6 weeks | 63.5 [58.0 to 68.9] | 66.6 [61.0 to 72.2]
  Kansas City Cardiomyopathy Questionnaire Overall Summary Score (KCCQ-OS) score - 12 weeks | 64.2 [58.8 to 69.6] | 61.7 [56.2 to 67.3]
  Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ-CS) score - 6 weeks | 66.6 [61.1 to 72.2] | 65.6 [60.0 to 71.3]
  Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ-CS) score - 12 weeks | 65.8 [60.3 to 71.2] | 60.2 [54.5 to 65.9]

8. Secondary Outcome: Proportion of Patients With a ≥ 5 Point Increase From Baseline in the Kansas City Cardiomyopathy Questionnaire Overall Summary Score (KCCQ-OS) at Either 6 Weeks or 12 Weeks of Follow-up Between Empagliflozin and Placebo.
Description: as for outcome 7
Time Frame: Baseline to Week 6 and Week 12
Population: The number of participants analyzed may differ from the overall number of participants analyzed due to missing data at certain timepoints for some participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 33 | 32
Participants
  KCCQ-OS score increase >/= 5 points (6 weeks): number analyzed (Participants) | 31 | 30
  KCCQ-OS score increase >/= 5 points (6 weeks) | 13 | 15
  KCCQ-OS score increase >/= 5 points (12 weeks): number analyzed (Participants) | 32 | 30
  KCCQ-OS score increase >/= 5 points (12 weeks) | 11 | 10
  KCCQ-CS score increase >/= 5 points (6 weeks): number analyzed (Participants) | 31 | 30
  KCCQ-CS score increase >/= 5 points (6 weeks) | 13 | 10
  KCCQ-CS score increase >/= 5 points (12 weeks): number analyzed (Participants) | 32 | 30
  KCCQ-CS score increase >/= 5 points (12 weeks) | 12 | 5

9. Secondary Outcome: Change in 6 Minute Walk Test From Baseline to Follow-up (Defined as Average of Measurements at 6 and 12 Weeks) Between Empagliflozin and Placebo.
Description: Change in 6 minute walk test from baseline to follow-up (defined as average of measurements at 6 and 12 weeks) between empagliflozin and placebo.
Time Frame: Baseline to Week 6 and Week 12
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 33 | 32
meters
  6-minute walk distance - 6 weeks | 202.5 [170.9 to 239.8] | 211.2 [177.0 to 252.0]
  6-minute walk distance - 12 weeks | 217.4 [183.3 to 257.9] | 174.7 [146.6 to 208.0]

10. Secondary Outcome: Change in N-terminal Pro B-type Natriuretic Peptide (NT-proBNP) From Baseline to Follow-up (Defined as Average of Measurements at 6 and 12 Weeks) Between Empagliflozin and Placebo.
Description: Change in N-terminal pro b-type natriuretic peptide (NT-proBNP) from baseline to follow-up (defined as average of measurements at 6 and 12 weeks) between empagliflozin and placebo.
Time Frame: Baseline to Week 6 and Week 12
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 33 | 32
pg/mL
  NT-proBNP - 6 weeks | 693 [556 to 865] | 655 [518 to 830]
  NT-proBNP - 12 weeks | 659 [528 to 822] | 802 [635 to 1013]

11. Secondary Outcome: Change in Brain Natriuretic Peptide (BNP) From Baseline to Follow-up (Defined as Average of Measurements at 6 and 12 Weeks) Between Empagliflozin and Placebo.
Description: Change in brain natriuretic peptide (BNP) from baseline to follow-up (defined as average of measurements at 6 and 12 weeks) between empagliflozin and placebo.
Time Frame: Baseline to Week 6 and Week 12
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 33 | 32
pg/mL
  BNP - 6 weeks | 143 [113 to 180] | 149 [116 to 191]
  BNP - 12 weeks | 144 [114 to 182] | 167 [130 to 214]

12. Secondary Outcome: Proportion of Patients With a ≥ 20% Decrease From Baseline in N-terminal Pro B-type Natriuretic Peptide (NT-proBNP) at Either 6 Weeks or 12 Weeks of Follow-up Between Empagliflozin and Placebo.
Description: Proportion of patients with a ≥ 20% decrease from baseline in N-terminal pro b-type natriuretic peptide (NT-proBNP) at either 6 weeks or 12 weeks of follow-up between empagliflozin and placebo.
Time Frame: Baseline to Week 6 and Week 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 33 | 32
Participants
  NT-proBNP decrease >/= 20% - 6 weeks: number analyzed (Participants) | 32 | 29
  NT-proBNP decrease >/= 20% - 6 weeks | 10 | 6
  NT-proBNP decrease >/= 20% - 12 weeks: number analyzed (Participants) | 32 | 30
  NT-proBNP decrease >/= 20% - 12 weeks | 11 | 2

13. Secondary Outcome: Proportion of Patients With a ≥ 20% Decrease From Baseline in Brain Natriuretic Peptide (BNP) at Either 6 Weeks or 12 Weeks of Follow-up Between Empagliflozin and Placebo.
Description: Proportion of patients with a ≥ 20% decrease from baseline in brain natriuretic peptide (BNP) at either 6 weeks or 12 weeks of follow-up between empagliflozin and placebo.
Time Frame: Baseline to Week 6 and Week 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 33 | 32
Participants
  BNP decrease >/= 20% - 6 weeks: number analyzed (Participants) | 32 | 30
  BNP decrease >/= 20% - 6 weeks | 12 | 6
  BNP decrease >/= 20% - 12 weeks: number analyzed (Participants) | 32 | 30
  BNP decrease >/= 20% - 12 weeks | 11 | 4

14. Secondary Outcome: Proportion of Patients With Both a ≥ 5 Point Increase From Baseline in KCCQ-OS and a ≥ 20% Decrease From Baseline in NT-proBNP at Either 6 Weeks or 12 Weeks of Follow-up Between Empagliflozin and Placebo.
Description: Proportion of patients with both a ≥ 5 point increase from baseline in Kansas City Cardiomyopathy Questionnaire Overall Summary Score (KCCQ-OS) and a ≥ 20% decrease from baseline in N-terminal pro b-type natriuretic peptide (NT-proBNP) at either 6 weeks or 12 weeks of follow-up between empagliflozin and placebo. The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a disease-specific health status instrument composed of 23 items that quantifies the domains of physical limitations, symptoms, self-efficacy, social limitation and quality of life from heart failure. Scores range from 0-100, in which higher scores reflect better health status. For the Kansas City Cardiomyopathy Questionnaire Overall Summary Score KCCQ-OS, a small but clinically meaningful change is considered to be ≥ 5 points.
Time Frame: Baseline to Week 6 and Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 32 | 30
Participants | 19 | 14

15. Secondary Outcome: Number of Participants With Diuretic Medication Adjustments During the Treatment Period Between Empagliflozin and Placebo
Description: Number of Participants with Diuretic Medication Adjustments During the Treatment Period Between Empagliflozin and Placebo
Time Frame: Baseline to Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 33 | 32
Participants
  Number of patients with no loop diuretic changes | 25 | 26
  Number of patients with loop diuretic changes | 8 | 6

16. Secondary Outcome: Change in Hemoglobin A1c From Baseline to Follow-up (Defined as Average of Measurements at 6 and 12 Weeks) Between Empagliflozin and Placebo.
Description: Change in Hemoglobin A1c from baseline to follow-up (defined as average of measurements at 6 and 12 weeks) between empagliflozin and placebo.
Time Frame: Baseline to Week 6 and Week 12
Measure: Mean (95% Confidence Interval); unit: percentage of hemoglobin
Arm/Group | Empagliflozin | Placebo
Number analyzed (Participants) | 33 | 32
percentage of hemoglobin
  Hemoglobin A1c - 6 weeks | 6.6 [6.3 to 6.9] | 6.5 [6.2 to 6.8]
  Hemoglobin A1c - 12 weeks | 6.8 [6.5 to 7.1] | 6.3 [6.1 to 6.6]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for up to 15 weeks. The adverse event collection period started at the time the patient signed consent at their Screening Visit, continued through a 12-week double-blind treatment period after randomization, and ended after completion of a 1-week follow-up period after completion of the double-blind treatment period.
Description: All adverse events were collected including Serious Adverse Events, Drug Adverse Events, Adverse Events of Special Interest and Urgent Outpatient Heart Failure Visits. A Drug Adverse Events is an adverse event which leads to premature and permanent discontinuation of study drug. Adverse Events of Special Interest include diabetic ketoacidosis, volume depletion, severe hypoglycemic events and non-traumatic lower limb amputations.
Arm/Group | Empagliflozin | Placebo
All-Cause Mortality (participants affected / at risk) | 1/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 8/33 | 9/32
Other Adverse Events (participants affected / at risk) | 19/33 | 16/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Empagliflozin (N=33) | Placebo (N=32)
Exacerbation of Heart Failure (Cardiac disorders) | 4 (4) | 4 (4)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Head Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Groin Abcess (Infections and infestations) | 1 (1) | 0 (0)
Hematuria (General disorders) | 1 (1) | 0 (0)
Hypotension (General disorders) | 1 (1) | 0 (0)
Osteoarthritis - left knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Volume Depletion (General disorders) | 1 (1) | 1 (1)
Worsening Tricuspid Valve Regurgitation (Cardiac disorders) | 1 (1) | 0 (0)
Endocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
CardioMEMS device recalibration (General disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Empagliflozin (N=33) | Placebo (N=32)
Acute Kidney Injury (General disorders) | 1 (1) | 2 (2)
Chest Pain (Cardiac disorders) | 2 (2) | 1 (1)
Cellulitis - bilateral legs (Infections and infestations) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Congestion (General disorders) | 1 (1) | 0 (0)
Contusion - scalp (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cough (General disorders) | 2 (2) | 0 (0)
Dysuria (General disorders) | 1 (1) | 0 (0)
Exacerbation of Heart Failure (Cardiac disorders) | 3 (3) | 3 (6)
Exertional Angina (Cardiac disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gout Flare (General disorders) | 1 (2) | 2 (2)
Hiccups (General disorders) | 1 (1) | 0 (0)
Asymptomatic hypoglycemia (Endocrine disorders) | 1 (1) | 1 (1)
Hypokalemia (General disorders) | 3 (4) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Increased craving for sweets (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Pulmonary Nodule (General disorders) | 1 (1) | 0 (0)
Quick Tempered (General disorders) | 1 (1) | 0 (0)
Abscess - bilateral - hips, buttocks and upper legs (Infections and infestations) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lower left extremity swelling (General disorders) | 1 (1) | 0 (0)
Vaginal Yeast Infection (Infections and infestations) | 1 (1) | 0 (0)
Vertigo (General disorders) | 1 (1) | 0 (0)
Volume Depletion (General disorders) | 3 (3) | 1 (1)
Worsening Gout (General disorders) | 1 (2) | 0 (0)
Wound Dehiscence (General disorders) | 1 (1) | 0 (0)
Bilateral Handshaking (General disorders) | 0 (0) | 1 (2)
Bloating (General disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Bursitis - left knee (General disorders) | 0 (0) | 1 (1)
Cerumen Impaction (General disorders) | 0 (0) | 1 (1)
Chest Discomfort (General disorders) | 0 (0) | 1 (2)
Decreased renal function (General disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (General disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (General disorders) | 0 (0) | 1 (2)
Dystrophic Toenails (General disorders) | 0 (0) | 1 (1)
Flu (General disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1)
Heart Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
ICD Battery Depletion (General disorders) | 0 (0) | 1 (1)
Indigestion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lightheadedness (General disorders) | 0 (0) | 1 (1)
Melena (General disorders) | 0 (0) | 1 (1)
Restrictive Ventilatory Defect (General disorders) | 0 (0) | 1 (1)
Sick Sinus Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Urinary Frequency (General disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (General disorders) | 0 (0) | 1 (2)
Worsening Edema (General disorders) | 0 (0) | 1 (1)
Worsening Urinary Urge Incontinence (General disorders) | 0 (0) | 1 (1)
Wrist Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Contusion - posterior lower left back (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Subsites will not publish until after all multicenter articles have been submitted for publication. Sponsor will have 18 months after the close of the Study at all sites to arrange for the submission of multicenter publications. If such multicenter publications are not submitted within 24 months after conclusion of the Study at all sites, Site Investigator and Subsite may publish the results from the Subsite's data, individually, pursuant to approval by Sponsor and Steering Committee.

DOCUMENTS (2):
  • Study Protocol (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT03030222/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT03030222/SAP_001.pdf